CLINICAL TRIAL: NCT05711667
Title: Letermovir Prophylaxis for Cytomegalovirus in Pediatric Hematopoietic Cell Transplantation
Brief Title: A Study of the Drug Letermovir as Prevention of Cytomegalovirus Infection After Stem Cell Transplant in Pediatric Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ACCL1932; NCI-2022-10769 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCL1932 (Other: Children's Oncology Group); COG-ACCL1932 (Other: DCP); ACCL1932 (Other: CTEP); U24CA196173 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2023-01-23; First posted 2023-02-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Specimen Handling; letermovir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARM A (Letermovir prophylaxis) (Experimental): Patients receive letermovir PO or IV over 60 minutes QD starting on day +1 post-transplant for 14 weeks. Patients undergo collection of blood samples for CMV PCR analysis weekly for 14 weeks, every 2 weeks until week 24, week 32, week 40 and week 52.
  Interventions: Procedure: Biospecimen Collection; Drug: Letermovir
- Arm B (No prophylaxis) (Active Comparator): Patients undergo collection of blood samples for CMV PCR analysis weekly for 14 weeks, every 2 weeks until week 24, week 32, week 40 and week 52. (CLOSED TO ACCURAL 09/29/2025)
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Letermovir — Given PO or IV
  Other Names: 2-((4S)-8-Fluoro-2-(4-(3-methoxyphenyl)piperazin-1-yl)-3-(2-methoxy-5-(trifluoromethyl)phenyl)-4H-quinazolin-4-yl)acetic Acid; AIC246; MK-8228; Prevymis
  Arms: ARM A (Letermovir prophylaxis)

SUMMARY:
This phase III single arm trial determines whether taking prophylactic letermovir will reduce the likelihood of infection with cytomegalovirus (CMV) in children and adolescents after stem cell transplant compared to estimated rate of infection without prophylaxis. The treatments used to prepare for HCT reduce the body's natural infection-fighting ability and increase the likelihood of an infection with a virus called cytomegalovirus. "Prophylaxis" means to take a drug to prevent a disease or side effect. Letermovir is an antiviral drug that stops cytomegalovirus from multiplying and may prevent cytomegalovirus infection and make the disease less severe.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of letermovir prophylaxis in the prevention of clinically significant CMV infection through Week 14 (~100 days) post-transplant in children and adolescents receiving allogeneic hematopoietic cell transplant (allo-HCT).

SECONDARY OBJECTIVE:

I. To evaluate the efficacy of letermovir prophylaxis as assessed by CMV-free survival through 24 weeks (~6 months) post-transplant in pediatric patients.

EXPLORATORY OBJECTIVES:

I. To evaluate the incidence of clinically significant CMV infection through 24 and 52 weeks post-transplant in patients who receive letermovir prophylaxis.

II. To evaluate overall survival post-transplant in patients who receive letermovir prophylaxis.

III. To evaluate time to engraftment and describe the cumulative incidence of non-engraftment among patients who receive letermovir.

IV. To examine the following clinically significant adverse events among patients exposed to letermovir: the total duration of neutropenia through week 14 (~100 days) post-transplant, the cumulative incidence of acute kidney injury and chronic kidney disease by 52 weeks post-transplant, and total inpatient hospital days by 14 weeks (~100 days) and 52 weeks post-transplant.

V. Describe patterns of anti-viral resistance at the onset of CMV DNAemia after allo-HCT among patients who receive letermovir prophylaxis.

VI. To describe immune reconstitution and CMV-specific immunity among patients who receive letermovir prophylaxis.

OUTLINE: Enrolled patients will be added to the single arm of the study and receive letermovir prophylaxis.

ARM A: Patients receive letermovir orally (PO) or intravenously (IV) over 60 minutes once daily (QD) starting on day +1 post-transplant for 14 weeks. Patients undergo collection of blood samples for CMV polymerase chain reaction (PCR) analysis weekly for 14 weeks, every 2 weeks until week 24, week 32, week 40 and week 52.

ARM B (CLOSED TO ACCRUAL 09/29/2025): Patients undergo collection of blood samples for CMV PCR analysis weekly for 14 weeks, every 2 weeks until week 24, week 32, week 40 and week 52.

ELIGIBILITY:
Inclusion Criteria:

* >= 2 years and < 18 years at the time of enrollment
* Weight must be >= 6 kg at the time of enrollment
* Planned allogeneic HCT (bone marrow, peripheral blood stem cell, or cord blood transplant)
* Patient must be CMV sero-positive (i.e., recipient CMV immunoglobulin G positive)

  * Note: If a patient has hypogammaglobulinemia but has previously been documented as CMV sero-positive, that is acceptable for study inclusion. For all patients already confirmed to be CMV IgG seropositive, repeat testing is not required within 7 days prior to enrollment. However, the laboratory data determining eligibility must be available in the patient's medical/research record for verification
* Patient is eligible for entry only if it is feasible for plasma CMV PCR testing to be sent and resulted within the protocol mandated time period

  * Reminder: To limit the likelihood of positive plasma CMV PCR post-enrollment and prior to start of study treatment period, it is recommended that patient enrollment proceed after patients start their transplant preparative regimen
* Patient must have a performance status corresponding to Lansky/Karnofsky scores > 50

  * Note: Use Lansky for patients =< 16 years of age and Karnofsky for patients > 16 years of age. For further reference, see performance status scales scoring under the standard sections for protocols among protocol reference materials provided on the Children's Oncology Group (COG) member website: https://members.childrensoncologygroup.org/prot/reference_materials.asp
* Estimated glomerular filtration rate > 10 mL/min/1.73 m^2 and not receiving dialysis
* Direct bilirubin =< 2 mg/dL and serum glutamate-pyruvate transaminase (SPGT) (alanine transaminase [ALT]) =<10 x upper limit of normal (ULN) for age

  * Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L

Exclusion Criteria:

* Expected inability to tolerate oral formulation of letermovir
* Hypersensitivity to letermovir or any component of the formulation
* History of CMV end organ disease within 6 months (180 days) prior to enrollment

  * Note: CMV end organ disease based on proposed definitions by Ljungman et al. and inclusive of proven, probable or possible disease
* Receipt of prior allogeneic HCT within one year of study enrollment
* Planned prophylactic administration of other anti-CMV medications or cellular products during the study, including:

  * High dose acyclovir (defined as doses >= 1500 mg/m^2 IV or >= 3200 mg oral (patients >= 40 kg) or >= 2400 mg/m^2 (patients < 40 kg) per day)
  * High dose valacyclovir (defined as doses >= 3000 mg/day in patients > 20 kg)
  * Foscarnet
  * Ganciclovir
  * Valganciclovir
  * CMV-directed cytotoxic T lymphocytes
* Planned receipt of the following contraindicated medications during the study treatment period; contraindicated medications must be discontinued at least 14 days prior to Day +1

  * Contraindicated medications for all patients:

    * Pimozide
    * Ergot alkaloids
  * Contraindicated medications for patients planned to receive cyclosporine:

    * Bosentan
    * Pitavastatin
    * Simvastatin
* Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted in certain animal reproduction studies with letermovir. A pregnancy test is required for female patients of childbearing potential
* Lactating females who plan to breastfeed their infants
* Sexually active female patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their letermovir treatment and through at least 4 weeks after the last dose of letermovir.

  * Note: No contraception measures are needed specifically during letermovir treatment for male trial participants who have pregnant or non-pregnant female partner(s) of reproductive potential. Contraception measures may be required for other aspects of the HCT procedure.
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinically significant cytomegalovirus (CMV) infection | Up to week 14 post-transplant
  Clinically significant CMV is defined as the first of (1) initiation of anti-CMV preemptive therapy for documented CMV DNAemia or (2) onset of CMV end-organ disease. Will estimate the cumulative incidence of clinically significant CMV at 14-weeks post-transplant and will report the corresponding 95% confidence interval.

SECONDARY OUTCOMES:
Detection of CMV DNAemia | Up to week 14 post-transplant
  Will estimate the cumulative incidence of CMV DNAemia at 14-weeks post-transplant by study arm and will report the corresponding 95% confidence intervals.
CMV-free survival | Up to 24 weeks post-transplant
  Will estimate the cumulative incidence of the occurrence of CMV DNAemia or death by week 24 post-transplant by study arm and will report the corresponding 95% confidence intervals.

OTHER OUTCOMES:
Clinically significant CMV infection in early follow up | Up to 24 weeks post-transplant
  Clinically significant CMV is defined as the first of (1) initiation of anti-CMV preemptive therapy for documented CMV DNAemia or (2) onset of CMV end-organ disease. Will estimate the cumulative incidence of clinically significant CMV at 24-weeks post-transplant and will report the corresponding 95% confidence interval.
Clinically significant CMV infection in late follow up | Up to 52 weeks post-transplant
  Clinically significant CMV is defined as the first of (1) initiation of anti-CMV preemptive therapy for documented CMV DNAemia or (2) onset of CMV end-organ disease. Will estimate the cumulative incidence of clinically significant CMV at 52-weeks post-transplant and will report the corresponding 95% confidence interval.
Overall survival (OS) in early follow up | Up to 24 weeks post-transplant
  The Kaplan-Meier method will be used to estimate the 24-week OS probability, as defined by time from transplant until death. The corresponding 95% confidence interval will be reported.
Overall survival (OS) in late follow up | Up to 52 weeks post-transplant
  The Kaplan-Meier method will be used to estimate the 52-week OS probability, as defined by time from transplant until death. The corresponding 95% confidence interval will be reported.
Neutrophil engraftment | Up to 60 days post-transplant
  Engraftment is defined as the first three days of neutrophil count values above 500 cells/μL. Will estimate the cumulative incidence of neutrophil engraftment at 60-days post-transplant and will report the corresponding 95% confidence interval.
Incidence of neutropenia | Up to 14 weeks post-transplant
  Neutropenia will be defined as an absolute neutrophil count < 500 cells/uL. Will estimate the median number of weeks of neutropenia post-transplant.
Incidence of acute kidney injury | Up to 52 weeks post-transplant
  Acute kidney injury will be defined as grade 3 or higher creatinine elevation using the common terminology criteria for adverse events (CTCAE) v5 definitions. Will estimate the cumulative incidence of acute kidney injury at 52-weeks post-transplant and will report the corresponding 95% confidence interval.
Incidence of chronic kidney disease | Up to 52 weeks post-transplant
  Chronic kidney disease will be defined as grade 2 or higher using the CTCAE v5 definitions. Will estimate the cumulative incidence of chronic kidney disease at 52-weeks post-transplant and will report the corresponding 95% confidence interval.
Number of inpatient hospital days | Up to 14 weeks post-transplant
  Will report the median number of inpatient hospital days post-transplant.
Number of inpatient hospital days | Up to one-year post-transplant
  Will report the median number of inpatient hospital days post-transplant.
Incidence of resistance to antiviral medications | Up to 14 weeks post-transplant
  Will estimate the cumulative incidence of resistance to antiviral medications among the patients who develop clinically significant CMV infection. This analysis will be restricted to patients with viral loads > 1000 IU/mL.
CD4+ lymphocyte count | At 14, 24, and 52 weeks post-transplant
  Will report the median CD4+ lymphocyte count.
CD8+ lymphocyte count | At 14, 24, and 52 weeks post-transplant
  Will report the median CD8+ lymphocyte count.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin W Elgarten, Principal Investigator — Children's Oncology Group
Locations (22):
- United States (22):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Children's Hospital of Michigan, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin